CLINICAL TRIAL: NCT00620178
Title: A REtrospective Study on the Effects of cAndesartan vs. Losartan on Blood Pressure, Health Care Consumption and cardiovascuLar Events In a "Real-liFe" GP sEtting in Sweden
Brief Title: Atacand (Candesartan) Real Life Study
Acronym: Real Life
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Anders Ljunggren, MD, AstraZeneca
Other Study IDs: NIS-CSE-ATA-2008/1
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: candesartan; losartan; blood pressure; cardiovascular disease; health care consumption
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — candesartan cilexetil; Losartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 1: Candesartan
  Interventions: Drug: Candesartan Cilexetil
- 2: Losartan
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Candesartan Cilexetil — oral once daily dose
  Other Names: ATACAND
  Groups: 1
Drug: Losartan — once daily oral dose
  Other Names: COZAAR
  Groups: 2

SUMMARY:
This study is a Swedish historical cohort study in patients prescribed Atacand or Cozaar for hypertension by selected primary care centres. Data will be extracted anonymously from electronic medical records. In addition, data regarding morbidity and mortality will be collected by merging the cohort with the following national registries: the Hospital Discharge Register (Slutenvårdsregistret), the Cause of Death Register and the Heart Intensive Care Admission (RIKS-HIA)

ELIGIBILITY:
Inclusion Criteria:

* Recorded blood pressure prior to therapy of > 140 and/or 90 mmHg
* Diagnosed as hypertensive within 15 months
* First prescription of Cozaar or Atacand between 1 January 1999 and 31 December 2007, inclusive

Exclusion Criteria:

* Previous prescription within 15 months any drug from the ATC groups C02, C03, C07 - C09 inclusive

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects are all patients found in EPS systems at the participating centres, who were prescribed candesartan (ATC-C09CA06) or losartan (C09CA01) for hypertension from 1 January 1999 - 31 December 2004 inclusive. The first found prescription is designated as index.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy objective is to investigate, on basis of 'first to event', the development of new cardiovascular diseases (CVD). | 1999 - 2007

SECONDARY OUTCOMES:
Cardiovascular disease states and procedures in the background and over the entire observation period will be identified by use of ICD-9 and ICD-10 coding for diseases of the cardiovascular system. Specifically are death, acute cardiovascular events, new | 1999 - 2007
Health care consumption will be assessed as contacts with health care providers, in-hospital time periods for cardiovascular disease states with associated therapeutic procedures, and times spent within various levels of care (e.g. ICU and general ward). | 1999 - 2007

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stålhammar, MD, Principal Investigator — Eriksbergs vårdcentral
Locations (1):
- Research Site, Uppsala, Sweden